CLINICAL TRIAL: NCT00351767
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Study to Assess the Effect of Topical Recombinant Human Vascular Endothelial Growth Factor (Telbermin) for Induction of Healing of Diabetic Foot Ulcers
Brief Title: A Study to Assess the Effect of Topical Recombinant Human Vascular Endothelial Growth Factor for Induction of Healing of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGF3554g
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Diabetes; Dabetic Feet
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: telbermin
- 2 (Experimental)
  Interventions: Drug: telbermin
- 3 (Experimental)
  Interventions: Drug: telbermin
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Topically applied
  Arms: 4
Drug: telbermin — Topically applied
  Arms: 1; 2; 3

SUMMARY:
This is a Phase II, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of three different doses of topically applied telbermin in subjects ≥ 18 years old with diabetic foot ulcers. Approximately 160 adult subjects with Type 1 or Type 2 diabetes mellitus will be enrolled at approximately 40 investigational sites in the United States and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to comply with the following: study drug gel application and dressing changes as instructed; use offloading footwear and practice of rubbing prevention (shear injury) of the study ulcer for the duration of the study; adherence to study requirements or use of adequate caregiver assistance
* For males and females of childbearing potential, use of an effective method of contraception
* Type 1 or 2 diabetes mellitus
* Inability to perceive 10 grams pressure in the peri-ulcer area using a Semmes-Weinstein 5.07 monofilament
* At least one full thickness (i.e., extending into the subcutaneous tissue or beyond) ulcer of the foot at or below the malleolus that does not involve bone, tendons, ligaments, or muscle (University of Texas Classification System for Diabetic Foot Wounds, Stage 1a)
* Estimated foot ulcer surface area, L x W, between ≥ 0.70 cm^2 and ≤ 5.0 cm^2 as measured at Treatment Day 1 Any subject who does not meet this criterion will not be eligible for randomization.
* Eye examination (indirect ophthalmoscopy, fundus photography, or fluorescein angiography) within 6 months prior to randomization with no indication of proliferative diabetic retinopathy or wet age-related macular degeneration

Exclusion Criteria:

* Presence of an active systemic or local cancer or tumor of any kind (with the exception of non-melanoma skin cancer)
* Proliferative diabetic retinopathy or wet age-related macular degeneration
* A history of pulmonary edema
* Active congestive heart failure
* Active infection or cellulitis of any ulcer on the study foot
* Active osteomyelitis of the study foot
* Active connective tissue disease
* Study ulcers with an etiology not related to diabetes (e.g., thermal, chemical, radiation insult)
* History of active Charcot foot of the study foot within 6 months of screening
* Treatment with systemic corticosteroids (equivalent to > 10 mg/day of prednisone) or immunosuppressive or chemotherapeutic agents within 14 days prior to the first study drug gel application or likelihood to receive one of these therapies during study participation
* Previous or current radiation therapy to the distal lower extremity or likelihood to receive this therapy during study participation
* Pregnancy or lactation
* Presence of more than two full-thickness ulcers on the study foot
* End-stage renal failure necessitating chronic hemodialysis or chronic ambulatory peritoneal dialysis
* Poor nutritional status
* Life expectancy of less than 3 years (in the opinion of the investigator)
* Known hypersensitivity to any ingredients of telbermin, placebo, or vehicle, including excipients in the formulation of telbermin or placebo gel
* Known prior inability to complete required study visits during study participation
* A psychiatric condition (e.g., suicidal ideation) or chronic alcohol or drug abuse problem, determined from the subject's medical history, which, in the opinion of the investigator, may pose a threat to subject compliance
* Use of a platelet-derived growth factor within the 28 days prior to screening
* Use of any investigational drug or therapy within the 28 days prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Skin re-epithelialization without drainage or dressing requirements | 12 weeks

SECONDARY OUTCOMES:
Complete closure of the study ulcer | 24 weeks
Durability of closure | Time to recurrence
Change and percent change in ulcer surface area | 12 and 24 weeks
Number of debridements performed | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pual Kwon, M.D., Study Director — Genentech, Inc.